CLINICAL TRIAL: NCT00691132
Title: Randomized Trial of PEITC as a Modifier of NNK Metabolism in Smokers
Brief Title: Phenethyl Isothiocyanate in Preventing Lung Cancer in Smokers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 2007NT127; R01CA122244 (NIH); 0712M22651 (Other: IRB, University of Minnesota)
Record Dates: First submitted 2008-06-04; First posted 2008-06-05 (Estimated); Results first posted 2017-04-04 (Actual); Last update posted 2017-05-12 (Actual); Status verified 2017-04

CONDITIONS: Lung Cancer; Tobacco Use Disorder
Keywords: non-small cell lung cancer; small cell lung cancer; tobacco use disorder
MeSH Terms: conditions — Lung Neoplasms; Tobacco Use Disorder; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma | interventions — phenethyl isothiocyanate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PEITC - Placebo (short-term trial) (Experimental): Participants are asked to smoke only deuterated NNK cigarettes (provided by the study) and record the exact number of cigarettes smoked and alcoholic drinks consumed each day for 1 month. Participants receive oral phenethyl isothiocyanate (PEITC) four times daily for 5 days in week 2 and oral placebo four times daily for 5 days in week 4. Participants keep a diary of all food and beverages consumed on the days that PEITC or placebo are taken.
  Interventions: Drug: phenethyl isothiocyanate; Other: placebo
- Placebo - PEITC (short-term trial) (Experimental): Participants receive oral placebo four times daily for 5 days in week 2 and oral PEITC four times daily for 5 days in week 4. Participants are also asked to smoke only deuterated NNK cigarettes, record the number of cigarettes smoked and alcoholic drinks consumed each day, and keep a food and beverage diary as in arm I.
  Interventions: Drug: phenethyl isothiocyanate; Other: placebo

INTERVENTIONS:
Drug: phenethyl isothiocyanate — Given orally
  Other Names: PEITC
Other: placebo — Given orally

SUMMARY:
RATIONALE: Chemoprevention is the use of certain drugs to keep cancer from forming. The use of phenethyl isothiocyanate may prevent lung cancer in people who smoke cigarettes.

PURPOSE: This randomized clinical trial is studying phenethyl isothiocyanate to see how well it works in preventing lung cancer in smokers.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine whether oral phenethyl isothiocyanate (PEITC) affects urinary levels of biomarkers of 4-(methylnitrosamino)-1-(3-pyridyl)-1-butanone (NNK) metabolism in current smokers.

Secondary

* To determine the effect of GSTM1 genotype on PEITC's impact on urinary biomarkers of NNK metabolism.
* To determine the effect of GSTM1 genotype on the metabolism and excretion of PEITC as measured by urinary levels of its major metabolite.
* To determine whether oral PEITC affects molecular markers of cell proliferation (Ki-67) and apoptosis (caspase-3 and TUNEL) in bronchial tissue.

OUTLINE: Patients are stratified according to GST genotypes (GSTM1 null-null genotype vs GSTM1-positive genotype). All participants are initially enrolled in the short-term trial. After the completion of the short-term trial, only those participants meeting certain criteria may proceed to the long-term trial.

* Short-term trial: Participants are randomized to 1 of 2 treatment arms.

  * Arm I: Participants are asked to smoke only deuterated NNK cigarettes (provided by the study) and record the exact number of cigarettes smoked and alcoholic drinks consumed each day for 1 month. Participants receive oral phenethyl isothiocyanate (PEITC) four times daily for 5 days in week 2 and oral placebo four times daily for 5 days in week 4. Participants keep a diary of all food and beverages consumed on the days that PEITC or placebo are taken.
  * Arm II: Participants receive oral placebo four times daily for 5 days in week 2 and oral PEITC four times daily for 5 days in week 4. Participants are also asked to smoke only deuterated NNK cigarettes, record the number of cigarettes smoked and alcoholic drinks consumed each day, and keep a food and beverage diary as in arm I.

After completion of the short-term trial, participants undergo a wash-out period for 1 month in which they are asked to resume smoking regular cigarettes. Participants are offered smoking cessation assistance, if desired. Only those participants meeting certain criteria may proceed to the long-term trial after the 1-month wash-out period.

* Long-term trial: Participants are randomized to 1 of 2 treatment arms.

  * Arm I: Participants receive oral PEITC twice daily for 12 months.
  * Arm II: Participants receive oral placebo twice daily for 12 months. Participants in both arms complete a 3-day food diary monthly for 12 months and a food-frequency questionnaire at baseline and at the completion of study treatment.

All participants undergo blood and urine sample collection periodically for laboratory studies. Participants enrolled in the long-term trial also undergo bronchoscopy and tissue biopsy at baseline and at the completion study treatment. Urine samples are examined by liquid chromatography-electrospray ionization-tandem mass spectrometry (LC-ESI-MS/MS) for various biomarkers. Tissue samples are examined by IHC for Ki-67, TUNEL, and caspase-3 expression.

ELIGIBILITY:
Inclusion criteria:

Initial from phone interview:

* Currently smoking 10-45 cigarettes per day for the past year;
* Between the ages of 21 and 70 years;
* In apparently good physical health with no unstable medical conditions including seizures or cancer;
* In stable and good mental health, i.e., currently do not experience unstable or untreated psychiatric diagnosis, including substance abuse, as determined by the DSM-IV criteria, during the past six months;
* Not using any other tobacco or nicotine-containing products;
* Not on methadone maintenance or stimulants such as ephedra; not a regular user of street drugs and if uses occasionally, willing to abstain during the study; not taking any drugs known to be P4501A6 substrates such as phenobarbital, rifampicin, dexamethasone, ketoconazole, methoxsalen, pilocarpine, or tranylcypromine due to their role in NNK metabolism;
* Does not average more than 21 alcoholic drinks per week;
* Willing to perform study activities such as having blood sample drawn, urine collection, multiple clinic visits;
* For female subjects of child bearing potential, not known to be pregnant or nursing, or planning to become pregnant within next 12 months.

For enrollment in the Short-Term Trial:

* Subjects who are generally healthy with liver enzyme and blood count values within the ranges shown below based on blood samples drawn at the second screening visit. Specifically:

  * White blood cells ≥ 3,000/mL
  * Total bilirubin ≤ 1.5 x upper limits of normal (ULN)
  * AST (SGOT)/ALT (SGPT) ≤ 2.5 x ULN
  * BUN and serum creatinine ≤ 1.5 x ULN

For enrollment in the Long-Term Trial:

* Participated in the short-term trial and invited to participate in the long-term trial;
* Possess the GSTM1 null-null genotype;
* Smoke 20 or more cigarettes/day with a cumulative smoking history of 20 or more pack-years (one pack-year equals to smoking a pack of cigarettes a day for one year);
* Normal liver enzymes based on blood sample drawn during 1 month wash-out;
* Determined to be a good candidate for the bronchoscopy procedure by a primary care physician.

Exclusion Criteria:

* Subjects with uncontrolled hypertension, uncontrolled diabetes mellitus, unstable coronary artery disease, history of cancer other than non-melanoma skin cancer, and pregnant or lactating women will not be eligible.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2009-02; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dorothy K. Hatsukami, PhD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Yuan JM, Stepanov I, Murphy SE, Wang R, Allen S, Jensen J, Strayer L, Adams-Haduch J, Upadhyaya P, Le C, Kurzer MS, Nelson HH, Yu MC, Hatsukami D, Hecht SS. Clinical Trial of 2-Phenethyl Isothiocyanate as an Inhibitor of Metabolic Activation of a Tobacco-Specific Lung Carcinogen in Cigarette Smokers. Cancer Prev Res (Phila). 2016 May;9(5):396-405. doi: 10.1158/1940-6207.CAPR-15-0380. Epub 2016 Mar 7. PMID 26951845
- [Derived] Dinh TN, Parat MO, Ong YS, Khaw KY. Anticancer activities of dietary benzyl isothiocyanate: A comprehensive review. Pharmacol Res. 2021 Jul;169:105666. doi: 10.1016/j.phrs.2021.105666. Epub 2021 May 12. PMID 33989764

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PEITC - Placebo (Short-term Trial) | Placebo - PEITC (Short-term Trial)
Started | 53 | 54 (107 total randomized. Approximately 1/2 per arm.)
Completed | 41 | 41 (45 completed, but 4 excluded b/c urinary measures indicated they did not smoke study cigarettes.)
Not Completed | 12 | 13
Not completed — Adverse Event | 2 | 3
Not completed — Withdrawal by Subject | 10 | 10

BASELINE CHARACTERISTICS:
Groups:
- Placebo - PEITC (Short-term Trial): Participants are asked to smoke only deuterated NNK cigarettes (provided by the study) and record the exact number of cigarettes smoked and alcoholic drinks consumed each day for 1 month. Participants receive oral placebo four times daily for 5 days in week 2 and oral PEITC four times daily for 5 days in week 4. Participants are also asked to smoke only deuterated NNK cigarettes, record the number of cigarettes smoked and alcoholic drinks consumed each day, and keep a food and beverage diary as in arm I.
  phenethyl isothiocyanate: Given orally
  placebo: Given orally
- Total: Total of all reporting groups
Arm/Group | PEITC - Placebo (Short-term Trial) | Placebo - PEITC (Short-term Trial) | Total
Number analyzed (Participants) | 41 | 41 | 82
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 41 | 41 | 82
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.9 (10.6) | 41.1 (9.6) | 41.0 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 21 | 38
  Male | 24 | 20 | 44
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 10 | 18
  White | 28 | 27 | 55
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 4 | 9
Region of Enrollment [Number; unit: participants]
  United States | 41 | 41 | 82
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 28.0 (4.8) | 28.0 (6.3) | 28.0 (5.6)
Level of Education [Number; unit: participants]
  High school or lower | 14 | 20 | 34
  College or higher | 27 | 21 | 48
Current smoking rate [Mean (Standard Deviation); unit: cigarettes/day] | 19.3 (6.6) | 19.0 (6.7) | 19.1 (6.6)
Cigarette smoking history [Mean (Standard Deviation); unit: years]
  Years of smoking | 14.7 (10.3) | 17.9 (9.4) | 16.3 (9.8)
  Age at starting smoking | 15.2 (4.9) | 15.1 (4.6) | 15.1 (4.7)
  Age became regular smokers | 18.6 (7.1) | 17.7 (5.2) | 18.1 (6.2)
Alcohol drinking [Number; unit: participants]
  Never | 14 | 17 | 31
  Monthly or less | 14 | 12 | 26
  Greater than monthly | 12 | 11 | 23
GSTM1 & GSTT1 genotypes [Number; unit: participants]
  Both present | 20 | 18 | 38
  Present/null | 3 | 4 | 7
  Null/present | 14 | 11 | 25
  Both null | 4 | 8 | 12

OUTCOME MEASURES:

1. Primary Outcome: Urinary Levels of Biomarkers of NNK Metabolism
Description: Urinary levels of Total ITC and PEITC-NAC by treatment sequence groups and treatment period.
Time Frame: 2 periods, 5 days each on PEITC or Placebo, with washout week between
Measure: Geometric Mean (95% Confidence Interval); unit: pmol/mg creatinine
Groups:
- PEITC-Placebo: Participants receive oral phenethyl isothiocyanate (PEITC) four times daily for 5 days in Period 1 and oral placebo four times daily for 5 days in Period 2, with washout period in between. Participants are asked to smoke only deuterated NNK cigarettes (provided by the study) and record the exact number of cigarettes smoked and alcoholic drinks consumed each day for 1 month.
- Placebo - PEITC: Participants receive oral placebo four times daily for 5 days in Period 1 and oral phenethyl isothiocyanate (PEITC) four times daily for 5 days in Period 2, with washout period in between. Participants are asked to smoke only deuterated NNK cigarettes (provided by the study) and record the exact number of cigarettes smoked and alcoholic drinks consumed each day for 1 month.
Arm/Group | PEITC-Placebo | Placebo - PEITC
Number analyzed (Participants) | 41 | 41
pmol/mg creatinine
  Period 1 - Total ITC | 42.8 [37.4 to 48.9] | 0.36 [0.19 to 0.54]
  Period 2 - Total ITC | 0.28 [0.13 to 0.46] | 49.7 [43.2 to 57.2]
  Period 1 - PEITC-NAC | 56.7 [46.3 to 69.3] | 0.27 [0.08 to 0.48]
  Period 2 - PEITC-NAC | 0.36 [0.01 to 0.85] | 68.1 [56.6 to 81.8]

2. Primary Outcome: Urinary Levels of Biomarkers of NNK Metabolism
Description: The ratio of urinary [pyridine-D4]hydroxy acid : total [pyridine-D4]NNAL will be measured. This ratio is not expected to be influenced by the number of cigarettes smoked per day, or smoking topography.
Time Frame: After 5 days of treatment
Measure: Geometric Mean (95% Confidence Interval); unit: pmol/mg creatinine
Groups:
- Placebo: Participants receive oral placebo four times daily for 5 days in either Period 1 or Period 2.
- PEITC: Participants receive oral phenethyl isothiocyanate (PEITC) four times daily for 5 days in either Period 1 or Period 2.
Arm/Group | Placebo | PEITC
Number analyzed (Participants) | 82 | 82
pmol/mg creatinine
  Total [pyridine-D4]NNAL | 0.366 [0.286 to 0.396] | 0.366 [0.285 to 0.396]
  [pyridine-D4]Hydroxy acid | 0.150 [0.128 to 0.175] | 0.140 [0.120 to 0.163]
  [pyridine-D4]Hydroxy acid :[pyridine-D4]total NNAL | 0.455 [0.409 to 0.508] | 0.420 [0.377 to 0.469]
Statistical Analysis 1: Comparison: Placebo vs PEITC; % difference between Placebo and PEITC periods in the ratio of [pyridine-D4]Hydroxy acid : [pyridine-D4] total NNAL; Test type: Superiority or Other; p = 0.023, Mixed Models Analysis; Mean Difference (Final Values) = -7.7, 95% CI 2-sided [-13.8 to -1.2]

3. Secondary Outcome: Effects of GSTM1 Genotype on Phenethyl Isothiocyanate (PEITC)-NNK Association and on the Metabolism and Excretion of PEITC
Description: Measured by high-performance liquid chromatography (HPLC). The aim is to determine the possible differential effects of GSTM1 genotype on PEITC excretion, using the method of Chung et al. The method will result in quantitative recovery of the PEITC-NAC.
Time Frame: After 5 days of PEITC treatment
Measure: Geometric Mean (95% Confidence Interval); unit: nmol/mg creatinine
Groups:
- GSTM1 Null: GSTM1 Null: gene for glutathione-S-transferase (GST) M1 (GSTM1), the homozygous deletion of the gene (GSTM1 null), leading to a lack of corresponding enzymatic activity.
- GSTM1 Present: GSTM1 Present: gene for glutathione-S-transferase (GST) M1 (GSTM1), present in one or both alleles, leading to a enzymatic activity.
Arm/Group | GSTM1 Null | GSTM1 Present
Number analyzed (Participants) | 37 | 45
nmol/mg creatinine
  PEITC-NAC | 71.7 [58.6 to 87.6] | 54.8 [45.6 to 65.8]
  Total ITC | 53.7 [46.7 to 61.8] | 40.5 [35.7 to 46.0]
Statistical Analysis 1: Comparison: GSTM1 Null vs GSTM1 Present; Total ITC; Test type: Superiority or Other; p = 0.005, ANOVA

4. Secondary Outcome: Effects of GSTT1 Genotype on Phenethyl Isothiocyanate (PEITC)-NNK Association and on the Metabolism and Excretion of PEITC
Description: Measured by high-performance liquid chromatography (HPLC). The aim is to determine the possible differential effects of GSTT1 genotype on PEITC excretion, using the method of Chung et al. The method will result in quantitative recovery of the PEITC-NAC.
Time Frame: After 5 days of treatment
Measure: Geometric Mean (95% Confidence Interval); unit: nmol/mg creatinine
Groups:
- GSTT1 Null: GSTT1 Null: gene for glutathione-S-transferase (GST) T1 (GSTT1), the homozygous deletion of the gene (GSTT1 null), leading to a lack of corresponding enzymatic activity.
- GSTT1 Present: GSTT1 Present: gene for glutathione-S-transferase (GST) T1 (GSTT1), present in one or both alleles, leading to a enzymatic activity.
Arm/Group | GSTT1 Null | GSTT1 Present
Number analyzed (Participants) | 19 | 63
nmol/mg creatinine
  PEITC-NAC | 67.1 [50.3 to 89.6] | 60.4 [51.5 to 70.7]
  Total ITC | 49.2 [40.0 to 60.4] | 45.1 [40.3 to 50.5]

5. Secondary Outcome: Combined Effects of GSTM1 and GSTT1 Genotype on Phenethyl Isothiocyanate (PEITC)-NNK Association and on the Metabolism and Excretion of PEITC
Time Frame: After 5 days of treatment
Measure: Geometric Mean (95% Confidence Interval); unit: nmol/mg creatinine
Groups:
- GSTM1 and GSTT1 Both Genes Null: GSTM1 & GSTT1 Null: genes for glutathione-S-transferase (GST) M1 & T1, the homozygous deletion of both genes (GSTM1 null and GSTT1 null), leading to a lack of corresponding enzymatic activity.
- GSTM1 and GSTT1 Only One Gene Present: GSTM1 or GSTT1 Present: at least one allele positive for either the gene for glutathione-S-transferase (GST) M1 or T1, but not or both genes, leading to moderate enzymatic activity.
- GSTM1 and GSTT1 Both Genes Present: GSTM1 and GSTT1 Present: at least one allele positive for both glutathione-S-transferase (GST) M1 and T1, leading to higher enzymatic activity.
Arm/Group | GSTM1 and GSTT1 Both Genes Null | GSTM1 and GSTT1 Only One Gene Present | GSTM1 and GSTT1 Both Genes Present
Number analyzed (Participants) | 12 | 32 | 38
nmol/mg creatinine
  PEITC-NAC | 85.4 [59.7 to 122.2] | 60.5 [48.6 to 75.3] | 56.9 [46.6 to 69.6]
  Total ITC | 59.6 [46.3 to 76.5] | 47.1 [40.4 to 55.0] | 41.5 [36.1 to 47.8]
Statistical Analysis 1: Comparison: GSTM1 and GSTT1 Both Genes Null vs GSTM1 and GSTT1 Only One Gene Present vs GSTM1 and GSTT1 Both Genes Present; Total ITC; Test type: Superiority or Other; p = 0.017, ANOVA

6. Secondary Outcome: Urinary Levels of [Pyridine-D4]Hydroxy Acid:Total [Pyridine-D4]NNAL Ratio by GSTM1 and GSTT1 Genotype.
Description: % Difference in ratio of urinary [pyridine-D4]hydroxy acid : total [pyridine-D4]NNAL while on PEITC compared to while on Placebo ((PEITC - Placebo) / PEITC) x 100%
Time Frame: After 5 days of treatment
Measure: Geometric Mean (95% Confidence Interval); unit: percentage of change in ratio
Arm/Group | GSTM1 and GSTT1 Both Genes Null | GSTM1 and GSTT1 Only One Gene Present | GSTM1 and GSTT1 Both Genes Present
Number analyzed (Participants) | 12 | 32 | 38
percentage of change in ratio | -15.6 [-26.7 to -2.9] | -3.1 [-14.6 to 9.9] | -9.4 [-17.4 to -0.6]
Statistical Analysis 1: Comparison: GSTM1 and GSTT1 Both Genes Null; Test type: Superiority or Other; p = 0.039, Mixed Models Analysis
Statistical Analysis 2: Comparison: GSTM1 and GSTT1 Only One Gene Present; Test type: Superiority or Other; p = 0.623, Mixed Models Analysis
Statistical Analysis 3: Comparison: GSTM1 and GSTT1 Both Genes Present; Test type: Superiority or Other; p = 0.045, Mixed Models Analysis

ADVERSE EVENTS:
Groups:
- Placebo (Short-term Trial): Participants are asked to smoke only deuterated NNK cigarettes (provided by the study) and record the exact number of cigarettes smoked and alcoholic drinks consumed each day for 1 month. Participants receive oral phenethyl isothiocyanate (PEITC) four times daily for 5 days in week 2 and oral placebo four times daily for 5 days in week 4. Participants keep a diary of all food and beverages consumed on the days that PEITC or placebo are taken.
  phenethyl isothiocyanate: Given orally
  placebo: Given orally
- Washout: 9 days between treatments
- PEITC (Short-term Trial): Participants receive oral placebo four times daily for 5 days in week 2 and oral PEITC four times daily for 5 days in week 4. Participants are also asked to smoke only deuterated NNK cigarettes, record the number of cigarettes smoked and alcoholic drinks consumed each day, and keep a food and beverage diary as in arm I.
  phenethyl isothiocyanate: Given orally
  placebo: Given orally
Arm/Group | Placebo (Short-term Trial) | Washout | PEITC (Short-term Trial)
Serious Adverse Events (participants affected / at risk) | 0/107 | 0/107 | 0/107
Other Adverse Events (participants affected / at risk) | 66/107 | 35/107 | 107/107
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (Short-term Trial) (N=107) | Washout (N=107) | PEITC (Short-term Trial) (N=107)
GI tract (Gastrointestinal disorders) | 30 (103) | 17 (35) | 62 (284) — Most common were dry mouth, taste alteration, stomachache, belching, flatulence, and diarrhea
Neurology (Nervous system disorders) | 17 (35) | 8 (11) | 25 (58)
Constitutional (General disorders) | 12 (24) | 6 (6) | 7 (13)
Other (General disorders) | 7 (14) | 5 (5) | 13 (24)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No